CLINICAL TRIAL: NCT00856505
Title: Everolimus and Mycophenolate Sodium as GvHD Prophylaxis in Allogeneic Stem Cell Transplantation
Brief Title: Safety Study of Calcineurin Inhibitor Free GvHD Prophylaxis in Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Prof. Jürgen Finke, University Hospital Freiburg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00557
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Hematologic Diseases
Keywords: Hematopoietic Stem Cell Transplantation; Drug Therapy, Combination; Immunosuppression
MeSH Terms: conditions — Hematologic Diseases | interventions — Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus and mycophenolate sodium (Experimental): Combination of experimental immunosuppressants for GvHD prophylaxis
  Interventions: Drug: Everolimus and mycophenolate sodium

INTERVENTIONS:
Drug: Everolimus and mycophenolate sodium — Everolimus tablets, 1.5mg/day bid, dosage adjusted to plasma levels Mycophenolate sodium, 720mg/day bid Duration: Mycophenolate tapering starts at day 56 after stem cell transplantation Everolimus tapering starts at day 100 after stem cell transplantation if no GvHD evident

SUMMARY:
In stem cell transplantation as treatment for malignant diseases, calcineurin inhibitors like cyclosporine A are commonly used to prevent tissue destruction (GvHD) by activated donor immune cells. The hypothesis for this study is, that replacing calcineurin inhibitors by everolimus and mycophenolate as GvHD prophylaxis not only reduces toxicity of the treatment but also improves tolerance induction of the donor T cells toward the host, eventually increasing the safety of stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hematologic malignancies, indicated for allogeneic stem cell transplantation:
* acute myeloid leukemia (AML), in CR1, ≥ CR2, primary refractory, relapse
* chronic myeloid leukemia (CML), in chronic phase, in acceleration or blast crisis
* myelodysplastic syndrome (MDS), RA/RARS (transfusion dependent), RAEB, RAEB-t and CMML
* Lymphoma:

  * plasmocytoma
  * immunocytoma (M. Waldenström)
  * chronic-lymphatic leukemia (CLL)
  * additional low and high grade Non-Hodgkin Lymphoma
* Hodgkins disease
* HLA-matched (HLA-A, -B, -DRB1) related or unrelated donor available
* Signed informed consent

Exclusion Criteria:

* CNS involvement by underlying disease
* Pulmonary disease with VC < 55%, DLCO < 40%
* Cardiac ejection fraction < 30%, uncontrollable arrhythmia
* Creatinin > 1,5 mg/dl or Creatinin-Clearance < 30 ml/min
* Bilirubin > 2 mg/dl
* Active Hepatitis B or C
* HIV serologic positive
* Pregnancy and lactation
* Pre-menstrual women without medical safe contraception
* Participation on another clinical trial in between 30 days before start or during the study only if the clinical trial interferes with the outcome measures.
* Known allergy to study medication or ingredients of the formulation
* Drug- or alcohol abuse
* Non-compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity according to CTCAE v3.0 | after 100 days and one year after treatment start

SECONDARY OUTCOMES:
Hematopoietic engraftment | day 30 after stem cell transplantation
Incidence of acute and chronic GvHD | one year after stem cell transplantation
Progression free survival | Day 100 and one year after stem cell transplantation
Overall survival | day 100 and one year after stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Finke, MD, Principal Investigator — University Medical Center Freiburg, Div. Hematology/Oncology; Reinhard Marks, MD, Study Director — University Medical Center Freiburg, Div. Hematology/Oncology
Locations (1):
- University Medical Center, Division Hematology/Oncology, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Schafer H, Blumel-Lehmann J, Ihorst G, Bertz H, Wasch R, Zeiser R, Finke J, Marks R. A prospective single-center study on CNI-free GVHD prophylaxis with everolimus plus mycophenolate mofetil in allogeneic HCT. Ann Hematol. 2021 Aug;100(8):2095-2103. doi: 10.1007/s00277-021-04487-y. Epub 2021 Mar 23. PMID 33755792